CLINICAL TRIAL: NCT03598010
Title: Safety, Tolerability and Preliminary Efficacy of Oral Administration of Tannins and Flavonoids in the Management of Pediatric Diarrhea
Brief Title: Safety, Tolerability and Preliminary Efficacy of Lenodiar Pediatric in Diarrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aboca Spa Societa' Agricola (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABO-LEN-02/19
Record Dates: First submitted 2018-07-02; First posted 2018-07-26 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Diarrhea; Chronic Diarrhea; Acute Diarrhea; Diarrhea, Infantile
MeSH Terms: conditions — Diarrhea; Diarrhea, Infantile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenodiar Pediatric in Acute/Prolonged Diarrhea (Experimental): LenoDiar Pediatric acts thanks to Actitan-F, a plant-based molecular complex resulting from Aboca research which reduces attacks of diarrhoea and normalises the consistency of stools, helping to rapidly restore a balanced intestinal function.
  Actitan-F counteracts the inflammation of the intestinal mucous membrane, always present in the case of diarrhoea, through two action mechanisms:
  * a protective action, achieved by forming a barrier-effect film to limit contact with microorganisms and irritants;
  * an antioxidant action on the free radicals which counteracts the irritation of the mucous membrane.
  Interventions: Device: Actitan-F (7dd)
- Lenodiar Pediatric in Chronic Diarrhea (Experimental): LenoDiar Pediatric acts thanks to Actitan-F, a plant-based molecular complex resulting from Aboca research which reduces attacks of diarrhoea and normalises the consistency of stools, helping to rapidly restore a balanced intestinal function.
  Actitan-F counteracts the inflammation of the intestinal mucous membrane, always present in the case of diarrhoea, through two action mechanisms:
  * a protective action, achieved by forming a barrier-effect film to limit contact with microorganisms and irritants;
  * an antioxidant action on the free radicals which counteracts the irritation of the mucous membrane.
  Interventions: Device: Actitan-F (28dd)

INTERVENTIONS:
Device: Actitan-F (7dd) — 1 sack every 4 hours, maximum 4 sacks/day for 7 days.
  Arms: Lenodiar Pediatric in Acute/Prolonged Diarrhea
Device: Actitan-F (28dd) — 1 sack every 4 hours, maximum 4 sacks/day for 28 days.
  Arms: Lenodiar Pediatric in Chronic Diarrhea

SUMMARY:
Evaluation of the efficacy of a treatment with Actitan-F, a natural molecular complex of tannins (from Agrimony and Tormentil) and flavonoids (Chamomile) in a pediatric population of children affected by acture/prolonged/chronic diarrhea

ELIGIBILITY:
Inclusion Criteria

1. Children of either sex aged between 1-12 years (inclusive);
2. Evidence of acute (onset <7 days prior to screening visit), prolonged (onset between 7 and 14 days prior to screening visit) or chronic (onset >14 days prior to screening visit) diarrhea.

   * Acute/Prolonged Diarrhea is defined as at least 3 evacuations of loose or watery stools (stools type 6-7 of Bristol scale) occurring in the 24 hours preceding the screening visit.
   * Chronic Diarrhea (>14 days duration), defined by passage of loose or watery stools (Bristol score 6 or 7) with or without an increase in frequency of bowel movements;
3. Evidence of mild to moderate dehydration, defined as a score 1-4 in the Clinical Dehydration Scale;
4. Parents/legal guardians availability to fill on a daily basis the electronic daily diary by a smartphone/tablet/laptop.
5. Parents/legal guardians* have given a written informed consent for participation in the study at the time of enrolment or before. The parent/legal guardian should also have agreed to bring the child for the visits scheduled in the protocol and to provide the requested information during the telephonic follow-up visit;
6. Parents/legal guardian able to understand the full nature and the purpose of the investigation, including possible risks and side effects, able to cooperate with the Investigator and to comply with the requirements of the entire investigation (ability to attend all the planned investigation visits according to the time limits included) based on Investigator's judgement.

Exclusion Criteria:

Exclusion Criteria

1. Children of female sex having started menarche;
2. Evidence of severe dehydration, defined as a score > 4 in the Clinical Dehydration Scale;
3. Known hypersensitivity to any of the components (active ingredients or excipients) of the investigational product;
4. Severely malnourished patients, defined as those patients with body weight < 50% for age;
5. History of immune diseases or conditions known to producing immunodeficiency (AIDS, other congenital immunodeficiency syndromes, anticancer drugs, etc.);
6. For acute/prolonged diarrhea only, patients who have received any of the following treatments within the 2 weeks before the screening/baseline visit:

   * Drugs with adsorbing properties, e.g. kaolin, pectin, bismuth subsalicylate;
   * Drugs that modify intestinal secretions, e.g. racecadotril;
   * Drugs that modify intestinal motility, e.g. opiates such as loperamide, atropine and other anti-cholinergic agents);
   * Laxatives
   * Antibiotics
7. History of seizures due to known or unknown causes;
8. Parents/legal guardians' refusal or inability to give written informed consent to participate in the study;
9. Parents/legal guardians who, in the opinion of the Investigator, are unable to fill up the electronic patient diary;
10. Patients who may not be possible to come for the scheduled visits;
11. Patients who have participated in any other clinical trial in the last 3 months prior to the start of the study.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Acute (onset <7 days) or Prolonged Diarrhea (onset ≥7 and ≤14 days): Response Rate (RR) measured after 4 treatment days. | Day0 to Day4
  Acute (onset <7 days) or Prolonged Diarrhea (onset ≥7 and <14 days): Response Rate (RR) measured after 4 treatment days. Patients will be considered as responders if they have experienced the passage of 2 formed stools or no stool for at least 12 consecutive hours during the 4 days treatment.
Chronic Diarrhea (onset >14 days): Response Rate (RR) measured across the whole treatment period | Day0 to Day28
  Chronic Diarrhea (onset >14 days): Response Rate (RR) measured across the whole treatment period (4 weeks). Patients will be considered as responders if they have experienced a 50% (or more) reduction in the number of days with at least 1 diarrheic stools (Bristol score 6 or 7) in the whole treatment period (4 weeks) compared to the 7 days prior the treatment (baseline).

SECONDARY OUTCOMES:
Number of episodes of daily watery evacuations | Day0-Day28
  Number of episodes of daily watery evacuations evaluated by means of the electronic patient diaries;
Number of unformed stools passed per 24-h interval, after the first dose | Day0-Day28
  Number of unformed stools passed per 24-h interval, after dosing evaluated by means of the electronic patient diaries
Number of treatment failures | Day0-Day28
  Number of treatment failures. A treatment failure is defined as clinical deterioration or worsening of symptoms or illness continuing after 120 h following the first dose evaluated by means of the electronic patient diaries
Difference in body weight | Day0-Day28
  Difference in body weight between baseline and End of Treatment
Frequency and severity of diarrhea associated symptoms | Day0-Day28
  Frequency and severity of diarrhea associated symptoms (nausea, vomiting, abdominal pain). Severity will be evaluated by means of a 0-4 Likert scale (0 = none; 1 = mild; 2 = moderate; 3 = severe; 4 = very severe);
Treatment Compliance | Day0-Day28
  Evaluation of the nr of sachets prescribed by the investigators and the % of compliance recorded
Proportion of patients requiring other (allowed) treatments | Day0-Day28
  Proportion of patients requiring other treatments in addition to Lenodiar Pediatric or to other concomitant treatments prescribed at baseline visit for diarrhea symptoms relief (e.g. parenteral rehydration and/or other medications) evaluated by means of the electronic patient diaries
Change in results of the Pediatric Quality of Life Questionnaire (PedsQL) | Day0-Day28
  Change in results of the Pediatric Quality of Life Questionnaire (PedsQL) between baseline and End of Treatment visits
Change in results in parent assessment of children Quality of Life (100 mm VAS) | Day0-Day28
  Change in results in parent assessment of children Quality of Life (100 mm VAS) between baseline and End of Treatment visits
Safety and tolerability of the treatment: Incidence of adverse events (AEs) and serious adverse events (SAEs), and rate of study discontinuations due to AEs/SAE; | Day0-Day28
  Incidence of adverse events (AEs) and serious adverse events (SAEs), and rate of study discontinuations due to AEs/SAE;

IPD SHARING:
Plan to Share IPD: No